CLINICAL TRIAL: NCT06757582
Title: Necrotizing Enterocolitis and Bowel Perforation in Very Preterm Infants - Long-term Follow up
Acronym: NOR-NEC
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/1976/REK nord
Record Dates: First submitted 2020-01-02; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Necrotizing Enterocolitis; Intestinal Perforation; Premature Infant Disease
Keywords: necrotizing enterocolitis; bowel perforation; preterm infant; long-term follow-up; quality of life
MeSH Terms: conditions — Enterocolitis, Necrotizing; Intestinal Perforation; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Hemoglobin, MCV, Hb-reticulocyte count, total reticulocytes, ferritin, cobalamine, albumin, calcium, phosphorous, blood urea nitrogen and creatinine + essential micronutrient (fat- and watersoluble vitamins)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Necrotizing enterocolitis (NEC) is a gastrointestinal syndrome characterized by transmural inflammation and necrosis of the large and/or small bowel and subsequent intramural gas-forming organisms into the intestinal wall. Some preterm infants also develop spontaneous intestinal perforations (SIP) without the classical bowel inflammation/necrosis seen in NEC. NEC and SIP can be challenging to differentiate. Severe cases of both conditions require surgery and often bowel resection, but mortality due to SIP seems lower.

Studies looking at "long-term prognosis" of infants with NEC and bowel perforation have mainly assessed outcome until 2-7 years of age. The primary school years is a vulnerable period for ex-preterm children. Disruption in learning and social integration is of great importance for their quality of life (QoL), but little data exist in this age group. Moreover, nutritional deficits (e.g. cobalamin- or iron-deficiency may impact cognitive development, but this has not been investigated in this "high-risk" population in school age. Authors of a recent systematic review on gastrointestinal sequel after NEC-surgery thus called for "more high-quality studies assessing long-term follow-up".

In this project we will study the long-term impact of surgery for NEC and bowel perforation in preterm infants, both with a quality of life (QoL) perspective and with a focus on development, growth, nutrition and persistent gastrointestinal problems.

DETAILED DESCRIPTION:
INTRODUCTION

Necrotizing enterocolitis (NEC) is a gastrointestinal syndrome characterized by transmural inflammation and necrosis of the large and/or small bowel and subsequent intramural gas-forming organisms into the intestinal wall. The incidence of NEC is inversely related to birth weight and gestational age (GA), with the majority of affected being very preterm infants (GA < 32 weeks), and in particular extremely preterm infants (GA < 28 weeks). In Scandinavia, the rates of NEC in extremely preterm infants is 6-9% (1-3). NEC is a devastating condition and one of the four main causes of mortality in neonatal intensive care units (NICUs) (4). Some preterm infants also develop spontaneous intestinal perforations (SIP) without the classical bowel inflammation/necrosis seen in NEC. NEC and SIP can be challenging to differentiate. Severe cases of both conditions require surgery and often bowel resection, but mortality due to SIP seems lower (5).

The clinical onset of NEC is usually in the second or third week of life. Typical symptoms and signs are a distended abdomen, periumbilical erythema, bloody stools, feeding intolerance and a generally unstable infant. However, the signs are non-specific, and the diagnosis is usually based on radiographic findings such as intramural bowel gas (6, 17, 18). The severity is classified by modified Bells criteria (18, 19). Stage I refers to suspected, but unconfirmed NEC. Stage II is radiographically confirmed NEC requiring medical therapy including broad-spectrum antibiotics and supportive care. Stage III patients demonstrate clinical signs of bowel necrosis, peritonitis, and septic shock, or radiographic findings of bowel perforation. These patients often receive surgery in addition to intensive care. The mortality rate of NEC is between 20-40%; highest in immature infants and/or stage III disease (20, 21).

Survivors of severe NEC (stage III) require long and often very intensive medical therapy that cause suffering for both patients and their families (18, 20). Moreover, medical therapy of patients with NEC requires huge resources for the neonatal unit and the health care system (20). Those who survive NEC have an increased risk of later gut-associated problems (e.g. short bowel syndrome and strictures) (18, 22), and neurodevelopmental disability (20, 23). Similar results have been observed in follow-up studies after SIP, but less data is available for this condition (23).

Although significant progress has been made in our understanding of NEC/SIP over the last decade, many questions remain regarding the long-term prognosis and optimal follow-up.

Studies looking at "long-term prognosis" of infants with NEC and bowel perforation have mainly assessed outcome until 2-7 years of age (20, 24). The primary school years is a vulnerable period for ex-preterm children. Disruption in learning and social integration is of great importance for their quality of life (QoL), but little data exist in this age group (25). Moreover, nutritional deficits (e.g. cobalamin- or iron-deficiency (26, 27) may impact cognitive development, but this has not been investigated in this "high-risk" population in school age. Authors of a recent systematic review on gastrointestinal sequel after NEC-surgery thus called for "more high-quality studies assessing long-term follow-up" (28).

In this project we will study the long-term impact of surgery for NEC and bowel perforation in preterm infants, both with a quality of life (QoL) perspective and with a focus on development, growth, nutrition and persistent gastrointestinal problems.

AIM

to collect long-term follow-up data on QoL, growth, development, biochemical nutritional status and persistent gastrointestinal symptoms among survivors of surgical NEC or bowel perforation in the neonatal period, in order to identify areas where we can improve or optimize follow-up.

RESEARCH QUESTION

What is the long-term outcome of preterm infants surviving surgical NEC or bowel perforation in the neonatal period?

ELIGIBILITY:
Inclusion Criteria:

* Case: All Norwegian very preterm infants (gestational age (GA) < 32 weeks) born during the 6-year period 2008-2013, diagnosed with surgical NEC or bowel perforation and surviving up to one year of age will be invited to participate as cases.
* Controls: For each case we will invite two controls matched for important clinical characteristics (e.g. sex, GA, clinical illness score, intracranial pathology, need for oxygen at discharge etc.).

Exclusion Criteria:

* not signing informed consent scheme

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Cases and Controls will be identified through the Norwegian Neonatal Network.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Pediatric quality of life (PedsQL) questionnaire | 2020-2021
  modular approach measuring health-related QoL in children and adolescents (2-18 years) incl. children with acute and chronic health conditions. This questionnaire comprises of 4 essential core domains namely: Physical Functioning, Emotional Functioning, Social Functioning and School Functioning.

SECONDARY OUTCOMES:
Pediatric quality of life (QoL) Gastrointestinal Symptoms | 2025
  Validated questionnaire assessing gastrointestinal problems.The questionnaire reports data on gastrointestinal symptoms, within 10 scales. The final score goes from 0-100 and higher values indicates less symptoms and better QoL.
5-15-R | 2025
  a standardized questionnaire for parents covering development and behavior of children and adolescents in ages 5 to 17 years
Blood samples | 2025
  Hb, leukocytes with differential count, platelets, reticulocytes, mean corpuscular volume, Hb in reticulocytes, ferritin, 25-OH vitamin D, cobalamine, urea, creatinine, calcium, phosphorous, 9 essential trace elements, a broad panel of other fat and water soluble vitamins.
  Data will be reported in SI units, or other conventional measures.
  For this outcome we will report data on number of participants with 1, 2, 3 or 4 or more abnormal laboratory values
Weight | 2025
  in kilogram and one decimal (e.g. 24.8 kg)
Height | 2025
  in cm
Head circumference | 2025
  in cm and one decimal (e.g. 45.7 cm)

CONTACTS AND LOCATIONS:
Overall Officials: Trond Flaegstad, MD, PhD, Study Director — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD for this study which is not a RCT

REFERENCES:
- [Background] Hau EM, Meyer SC, Berger S, Goutaki M, Kordasz M, Kessler U. Gastrointestinal sequelae after surgery for necrotising enterocolitis: a systematic review and meta-analysis. Arch Dis Child Fetal Neonatal Ed. 2019 May;104(3):F265-F273. doi: 10.1136/archdischild-2017-314435. Epub 2018 Jun 26. PMID 29945925
- [Result] Neu J. Necrotizing enterocolitis: the mystery goes on. Neonatology. 2014;106(4):289-95. doi: 10.1159/000365130. Epub 2014 Aug 20. PMID 25171544